CLINICAL TRIAL: NCT05287139
Title: Quality of Life of Women With Hormone Receptor-Positive Metastatic Breast Cancer Treated in the First-line Setting: Comparison Between Public and Private Institutions.
Brief Title: QOL of Women With HR-Positive Metastatic BC Treated in the First-line Setting: Comparison Between Public and Private Institutions.
Acronym: BRAVE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Principal Investigator, Debora de Melo Gagliato Jardim, MD, Beneficência Portuguesa de São Paulo
Other Study IDs: BRAVE
Record Dates: First submitted 2022-03-10; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Quality of Life; Breast Neoplasm Female
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospital Beneficência Portuguesa de SP - BP1: Patients from private institutions.
  Interventions: Other: Quality of Life
- Hospital Pérola Byington - HPB2: Patients from public institutions.
  Interventions: Other: Quality of Life

INTERVENTIONS:
Other: Quality of Life — Assessment of patients' quality of life using the EORTC QLQ-C30 and EORTC-QLQ-BR 23 questionnaires

SUMMARY:
Assess the quality of life in patients with hormone receptor positive, human epidermal growth factor receptor-type 2 negative metastatic breast cancer treated in first line (patients with new metastasis or recurrence during adjuvant endocrine therapy): comparison between public and private institutions. The hypothesis to be evaluated is that patients treated in private institutions have a better quality of life when compared to patients treated in public institutions.

DETAILED DESCRIPTION:
The main objective of the study is to assess the quality of life using the EORTC-QLQ-C30 (EORTC Quality of Life Questionnaire) and the EORTC-QLQ-BR23 (EORTC Quality of Life Questionnaire - Breast Cancer) of a patient with metastatic breast cancer hormone receptor positive human epidermal growth factor receptor-type 2 negative receiving treatment in the first-line scenario, comparing public and private institutions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate by signing a document of free and informed consent (ICF), indicating that the research participant was informed about all relevant aspects of the study;
* Female patients ≥ 18 years of age;
* Patients diagnosed with hormone receptor positive, human epidermal growth factor receptor-type 2 -negative metastatic breast cancer; in first-line treatment (metastatic de novo disease or patients with recurrence during adjuvant endocrine therapy).
* First-line treatment can be considered as cytotoxic chemotherapy, isolated endocrine therapy or endocrine therapy in combination with 4/6 cyclin inhibitors.
* Patients on treatment for at least three (3) months and no more than eighteen (18) months.
* Have performance status Eastern Cooperative Oncology Group (ECOG scale) of 0-2.
* Do not present other concomitant neoplasms.

Exclusion Criteria:

* Patients who refuse to participate.
* Illiterate patients, with low levels of education or cognitive deficits that make it difficult to answer the questions of the data collection instrument.
* Patients with life expectancy <3 months.
* Treatment with any product under investigation during the last 28 days.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at the oncology outpatient clinic of Hospital Beneficência Portuguesa in São Paulo and Hospital Perola Byington
Sampling Method: Non-Probability Sample
Enrollment: 202 (Estimated)
Dates: Start 2021-07-14 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Assess the quality of life | Baseline
  Assess the quality of life using the EORTC-QLQ-C30 (EORTC Quality of Life Questionnaire)
Assess the quality of life in breast cancer | Baseline
  Assess the quality of life using the EORTC-QLQ-BR 23 (EORTC Quality of Life Questionnaire - Breast Cancer).

CONTACTS AND LOCATIONS:
Overall Officials: Débora G Jardim, MD, Principal Investigator — Beneficência Portuguesa de São Paulo
Locations (1):
- Hospital Pérola Byington, São Paulo, Brazil